CLINICAL TRIAL: NCT02864433
Title: Evaluation of a Pilot Program to Introduce Cholera Vaccine in Haiti as Part of Global Cholera Control Efforts
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Partners in Health (Other); Harvard Medical School (HMS and HSDM) (Other); Massachusetts General Hospital (Other); Ministry of Health, Haiti (Unknown)
Responsible Party: Principal Investigator, Louise Ivers, MD, Associate Physician, Brigham and Women's Hospital
Other Study IDs: 2012P000393; R01AI099243 (NIH)
Record Dates: First submitted 2014-05-19; First posted 2016-08-12 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Cholera; Diarrhea
Keywords: cholera; oral cholera vaccine; diarrhea
MeSH Terms: conditions — Cholera; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples from patients with acute watery diarrhea were collected and tested for cholera by rapid test and also by culture.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Controls for non-cholera diarrhea cases: - Community members that did not have diarrhea between date of study commencement, and time of presentation of the case
- Non-cholera diarrhea cases: - Cases of acute watery diarrhea that present for healthcare at the study sites, but that test negative for cholera
- Controls for cholera cases: - Community members that did not have diarrhea between date of study commencement, and time of presentation of the case
- Cholera cases: - Those with cholera-related diarrhea who present to healthcare at the study sites.

SUMMARY:
The investigators aim to evaluated a public health program in Haiti that introduced an oral cholera vaccine as part of comprehensive control efforts for a major cholera epidemic. Although the vaccine (Shanchol(R)) had been demonstrated to be very safe, and effective at preventing cholera in many settings, it had not extensively been used to control an outbreak, and it had not been extensively studied in populations that were previously naive to cholera (i.e. countries that had never had cholera before). This cholera epidemic was the first ever report of cholera in Haiti.

After the cholera vaccination campaign was complete, the investigators aimed to evaluate the field efficacy of the vaccination campaign by evaluating the number of cases of cholera, and determining if cholera patients had been vaccinated. The investigators compared the rate of vaccination in cholera cases to controls from the community that had not had cholera in a case-control study.

The investigators also performed a second study - a bias-indicator study - that enrolled patients with non-cholera diarrhea, and community controls. The role of the bias-indicator study was to evaluate for potential sources of bias, since the investigators could expect that cholera vaccination should have no effect on non-cholera diarrhea.

ELIGIBILITY:
Inclusion criteria for cholera cases:

* Seeks treatment for acute non-bloody diarrhea (defined as 3 or more loose, watery or liquid stools in a 24-hour period with an onset of 3 days or fewer prior to presentation) at a participating study site
* Diarrhea episode is diagnosed as cholera, confirmed by Crystal VC rapid test and culture
* Resident of Bocozel or Grande Saline at the time of study initiation
* Was eligible for the vaccination campaign (i.e. ≥ 12 months of age at the time of completion of the vaccine campaign, not pregnant during the vaccination campaign).

Exclusion criteria for cholera cases:

* < 12 months of age at the time of completion of the cholera vaccine campaign
* Pregnant at the time of the vaccination campaign

Inclusion criteria for non-cholera diarrhea cases:

* Seeks treatment for acute non-bloody diarrhea (as defined above) at a participating study site
* Culture negative cholera by Crystal VC rapid test and culture
* Resident of Bocozel or Grande Saline at the time of study initiation
* Was eligible for the vaccination campaign (≥ 12 months of age at the time of completion of the vaccine campaign, not pregnant at the time of the campaign)

Exclusion criteria for non-cholera diarrhea cases:

* < 12 months of age at the time of completion of the cholera vaccine campaign
* Pregnant at the time of the vaccination campaign

Inclusion criteria for all controls:

* Did not seek treatment for diarrhea between the date that study enrollment began and corresponding case's symptom onset (defined below)
* Resident of Bocozel or Grande Saline at the time of study initiation
* Was eligible for the vaccination campaign (≥ 12 months of age at the time of completion of the vaccine campaign, not pregnant at the time of the vaccination campaign)

Exclusion criteria for cholera controls and secondary controls:

* < 12 months of age at the time of completion of the cholera vaccine campaign
* Pregnant at the time of completion of the cholera vaccine campaign

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in the catchment area of the vaccine campaign, in the rural regions of Bocozel and Grande Saline, located in the Artibonite Department of Haiti. Bocozel has a catchment population of approximately 56,000 people and Grande Saline has a catchment population of approximately 21,000 people. These two neighboring sections are one of two Haitian locations in which the two-dose Shanchol oral cholera vaccine will be implemented as part of the vaccination campaign in 2012. Key stakeholder meetings conducted by PIH staff among diverse groups of community members in Bocozel suggest broad acceptance of the vaccine. Based on these meetings and reported oral cholera vaccine uptake in other countries, we estimate that vaccine uptake will be 80% or higher in Bocozel.
Sampling Method: Non-Probability Sample
Enrollment: 2207 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
cholera-related diarrhea | We will report diarrhea rates at 12 months after the cholera vaccination campaign
  Diarrhea will be determined by clinical symptoms of acute watery diarrhea (3 stools in the past 24 hours).
  'Cholera' designation will be determined by rapid test and confirmed by bacteriologic culture.
cholera-related diarrhea | We will report diarrhea rates at 24 after the cholera vaccination campaign
  Diarrhea will be determined by clinical symptoms of acute watery diarrhea (3 stools in the past 24 hours).
  'Cholera' designation will be determined by rapid test and confirmed by bacteriologic culture.
cholera-related diarrhea | We will report diarrhea rates at 60 months after the cholera vaccination campaign
  Diarrhea will be determined by clinical symptoms of acute watery diarrhea (3 stools in the past 24 hours).
  'Cholera' designation will be determined by rapid test and confirmed by bacteriologic culture.

SECONDARY OUTCOMES:
non-cholera diarrhea | We will report diarrhea rates at 12 months after the cholera vaccination campaign
  Diarrhea will be determined by clinical criteria for acute watery diarrhea (3 stools in the past 24 hours).
  'Non-cholera' designation will be determined by rapid test for cholera and bacteriologic culture (negative rapid test, culture negative = 'non-cholera')
non-cholera diarrhea | We will report diarrhea rates at 24 months after the cholera vaccination campaign
  Diarrhea will be determined by clinical criteria for acute watery diarrhea (3 stools in the past 24 hours).
  'Non-cholera' designation will be determined by rapid test for cholera and bacteriologic culture (negative rapid test, culture negative = 'non-cholera')
non-cholera diarrhea | We will report diarrhea rates at 60 months after the cholera vaccination campaign
  Diarrhea will be determined by clinical criteria for acute watery diarrhea (3 stools in the past 24 hours).
  'Non-cholera' designation will be determined by rapid test for cholera and bacteriologic culture (negative rapid test, culture negative = 'non-cholera')

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Ivers, MB,BCh,BAO, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Hopital St Nicholas, Saint-Marc, Haiti